CLINICAL TRIAL: NCT02962739
Title: The Cellular Pharmacology of F-TAF in Dried Blood Spots
Acronym: TAF-DBS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16-0972
Record Dates: First submitted 2016-11-08; First posted 2016-11-11 (Estimated); Results first posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Healthy Volunteers
Keywords: healthy volunteers
MeSH Terms: interventions — Emtricitabine; tenofovir alafenamide; emtricitabine tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 33%/67% dosing (Active Comparator): The 33% and 67% dosing regimens will use skipped doses spaced by days (i.e. 67% is two daily doses followed by skipping a day, repeated for 12 weeks; 33% dosing is a daily dose followed by two skipped days, repeated for 12 weeks).
  Interventions: Drug: emtricitabine 200 mg/tenofovir alafenamide 25mg
- 33%/100% dosing (Active Comparator): The 33% dosing regimens will use skipped doses spaced by days (i.e. 33% dosing is a daily dose followed by two skipped days, repeated for 12 weeks). 100% will dose daily for 12 weeks, no skipped doses.
  Interventions: Drug: emtricitabine 200 mg/tenofovir alafenamide 25mg
- 67%/33% dosing (Active Comparator): The 33% and 67% dosing regimens will use skipped doses spaced by days (i.e. 67% is two daily doses followed by skipping a day, repeated for 12 weeks; 33% dosing is a daily dose followed by two skipped days, repeated for 12 weeks).
  Interventions: Drug: emtricitabine 200 mg/tenofovir alafenamide 25mg
- 67%/100% dosing (Active Comparator): 67% dosing regimens will use skipped doses spaced by days (i.e. 67% is two daily doses followed by skipping a day, repeated for 12 weeks. 100% will dose daily for 12 weeks, no skipped doses.
  Interventions: Drug: emtricitabine 200 mg/tenofovir alafenamide 25mg
- 100%/33% dosing (Active Comparator): The 33% dosing regimens will use skipped doses spaced by days (i.e. 33% dosing is a daily dose followed by two skipped days, repeated for 12 weeks). 100% will dose daily for 12 weeks, no skipped doses.
  Interventions: Drug: emtricitabine 200 mg/tenofovir alafenamide 25mg
- 100%/67% dosing (Active Comparator): 67% dosing regimens will use skipped doses spaced by days (i.e. 67% is two daily doses followed by skipping a day, repeated for 12 weeks. 100% will dose daily for 12 weeks, no skipped doses.
  Interventions: Drug: emtricitabine 200 mg/tenofovir alafenamide 25mg

INTERVENTIONS:
Drug: emtricitabine 200 mg/tenofovir alafenamide 25mg — 1 tablet of Descovy contains emtricitabine 200 mg/tenofovir alafenamide 25mg
  Other Names: Descovy

SUMMARY:
Adherence to daily dosing is very important for how well Emtricitabine/Tenofovir Alafenamide (F/TAF) works for treatment of chronic human immunodeficiency virus (HIV), or prevention of HIV acquisition. Methods to measure medication adherence to Tenofovir disoproxil fumarate (tenofovir DF, TDF), a similar but different prodrug of tenofovir, have been developed but cannot be extrapolated to F-TAF. By measuring F-TAF (the drug) and metabolites in the blood cells and dried blood spots, the study plans to see if these results predict adherence to taking the drug. The goal of this study is to vary the amount of F-TAF dosing and see if the drug levels in dried blood spots (DBS) change in a predictable way. This study will mimic different levels of adherence (33%, 67%, and 100% of daily dosing) using directly observed therapy (DOT) to establish the relationship between F-TAF in dried blood spots and adherence. Investigators will also measure drug in hair clippings to see if hair or DBS are a better predictor of adherence.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory 18-59 year old adults. Enrollment will proceed without the need to meet specific race/gender targets, but balanced gender and African-Americans and Latino representation will be sought.
2. Ability to comply with study procedures, including directly observed dosing visits and availability and use of video streaming technology.

Exclusion Criteria:

1. Inability to give informed consent
2. Pregnancy or plan to become pregnant in the next 12 months or unwillingness to use birth control
3. Current breastfeeding
4. High risk of HIV-1 infection, for example:

   * sexually active with an HIV infected partner;
   * men who have sex with men who may engage in condomless intercourse with HIVinfected partners, or
   * partner of unknown status during the study;
   * males or females who exchange sex for money, shelter, or gifts;
   * active injection drug use or during the last 12 months;
   * newly diagnosed sexually transmitted infections in last 6 months
5. Positive screening HIV+ ELISA or suspected acute HIV infection in the opinion of the clinician. Example signs and symptoms of acute HIV infection include combinations of:

   * fever,
   * headache,
   * fatigue,
   * arthralgia,
   * vomiting,
   * myalgia, .
   * diarrhea,
   * pharyngitis,
   * rash,
   * night sweats, and
   * adenopathy (cervical or inguinal)
6. Positive Hepatitis B Virus (HBV) surface antigen test at screening
7. Active psychiatric illness, social condition, or alcohol/drug abuse that, in the opinion of the investigators, would interfere with study requirements.
8. Glomerular Filtration Rate (GFR) estimate < 60 ml/min (MDRD equation).
9. Urine dipstick protein ≥ 2+
10. Total bilirubin and/or hepatic transaminases (ALT and AST) ≥ 2.5x upper limit of normal
11. Absolute neutrophil count ≤ 1,500/mm3, platelets count ≤ 100,000/mm3, or hemoglobin ≤ 10 g/dL.
12. Symptomatic hemoglobinopathies or active hemolysis.
13. History of pathological, non-traumatic bone fractures
14. Any laboratory value or uncontrolled medical conditions that, in the opinion of the investigators, would interfere with the study conditions such as, heart disease and/or cancer.
15. Prohibited concomitant medications are:

    * investigational agents (within 30 days of enrollment),
    * aminoglycosides,
    * ganciclovir/valganciclovir,
    * chronic high-dose acyclovir/valacyclovir (>800mg acyclovir or > 500mg valacyclovir for 7 days),
    * cyclosporine, amphotericin B, foscarnet, and cidofovir, and products with same or similar active ingredients as the study medications including TRUVADA®, ATRIPLA®, COMPLERA®, EMTRIVA®, VIREAD®; or drugs containing lamivudine or adefovir, which are close analogs of FTC and tenofovir, respectively.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Anderson, PharmD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado- Anschutz Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yager J, Castillo-Mancilla J, Ibrahim ME, Brooks KM, McHugh C, Morrow M, McCallister S, Bushman LR, MaWhinney S, Kiser JJ, Anderson PL. Intracellular Tenofovir-Diphosphate and Emtricitabine-Triphosphate in Dried Blood Spots Following Tenofovir Alafenamide: The TAF-DBS Study. J Acquir Immune Defic Syndr. 2020 Jul 1;84(3):323-330. doi: 10.1097/QAI.0000000000002354. PMID 32539288

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 33%/67% Dosing | 33%/100% Dosing | 67%/33% Dosing | 67%/100% Dosing | 100%/33% Dosing | 100%/67% Dosing
Started | 6 | 7 | 7 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 5 | 6
Not Completed | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are not stratified based on dosing regimen. Dosing Arms were combined, regardless of dosing regimen order (i.e. all 33%, regardless if 33% regimen followed by other regimen (100% or 67%), or other regimen (100% or 67%) followed by 33%) to be consistent with data collection, protocol subject randomization and journal publications. Combined arms best categorize the study, population, and data.
Groups:
- All Dosing Regimens: Baseline characteristics for all 35 subjects analyzed. Baseline characteristics not stratified based on dosing regimen. Arms were combined to be consistent with protocol subject randomization. Subjects were randomized to one of six arms. Combined arms best categorize the study, population, and data.
Arm/Group | All Dosing Regimens
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants] — Population: 3 subjects withdrew- only 35 of 38 enrolled were analyzed
  Participants
    <=18 years | 0
    Between 18 and 65 years | 35
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 3 subjects withdrew- only 35 of 38 enrolled were analyzed.
  Participants
    Female | 17
    Male | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 38 subjects started study procedures. Of 38, 3 withdrew thus only 35 were analyzed.
  Participants
    African American | 5
    Caucasian | 24
    Hispanic | 6

OUTCOME MEASURES:

1. Primary Outcome: Steady State Concentrations of TFV-DP for Different Dosing Patterns of Descovy
Description: Tenofovir diphosphate (TFV-DP) concentrations in dried blood spots (DBS) respective to dosing regimens of 33%, 67%, 100% of daily dosing.
Time Frame: Assessed weekly for 9 months
Population: 34 participants received 2 of 3 dosing regimens and 1 participant only completed through week 8 of the second regimen, resulting in a total of 69 observations.
Measure: Mean (Standard Deviation); unit: fmol/punch
Groups:
- DOT 33%: 33% of daily dosing; dosing on day one followed by skipped doses on days two and three, repeated for 12 weeks
- DOT 67%: 67% of daily dosing; dosing on days one and two, skipped dose on day three, repeated for 12 weeks
- DOT 100%: 100% of daily dosing:dosing every day for 12 weeks
Arm/Group | DOT 33% | DOT 67% | DOT 100%
Number analyzed (Participants) | 23 | 23 | 23
fmol/punch | 657 (186) | 1451 (501) | 2381 (601)

ADVERSE EVENTS:
Time Frame: Time of consenting to study exit (Week 36 or earlier), Max 10 months.
Description: AEs were graded per the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.0, November, 2014. Available: http://rsc.tech-res.com/safetyandpharmacovigilance/.
  Arms were combined as Descovy was FDA approved for daily use (100% dosing) at the time of study initiation- no arm was considered to be more at risk for AEs than another.
Groups:
- All Subjects: At study initiation Descovy was FDA approved for daily dosing (100% daily dosing). Thus, the AE profile was already established for 100% dosing and AE rates in the lower doses (33% and 67%) would not exceed the established rate for daily dosing (100%). This study was not designed to collect new safety data or to update the established AE/Safety profiles for Descovy. Therefore AE data was combined for all dosing regimens.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 2/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=38)
traumatic leg fracture (Injury, poisoning and procedural complications) | 1 (1) — traumatic leg fracture unrelated to study drug
Pleurisy VS costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) — Left-sided chest pain, pain was exertional and with movement. ED ruled out PE and cardiac issues, and thought it was muscular and potentially "inflammatory" in etiology. Pain resolved and no reason to believe related to study procedures.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=38)
Abnormal Labs (General disorders) | 15 (29)
Cold Symptoms (General disorders) | 31 (62)
Diarrhea (Gastrointestinal disorders) | 10 (14)
Abdominal Pain (Gastrointestinal disorders) | 4 (5)
Headache (General disorders) | 8 (14)
Nausea (Gastrointestinal disorders) | 18 (22)
Vomiting (Gastrointestinal disorders) | 10 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT02962739/Prot_SAP_000.pdf